CLINICAL TRIAL: NCT00112866
Title: Phase II Trial of EMD 121974 for Recurrent Glioblastoma: A Clinical Trial With Tissue Correlates of Response
Brief Title: Cilengitide in Treating Patients Who Are Undergoing Surgery for Recurrent or Progressive Glioblastoma Multiforme
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: due to poor accrual
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02653; NCI-2012-02653 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000428409; NABTC-03-02 (Other: North American Brain Tumor Consortium); NABTC-03-02 (Other: CTEP); U01CA062399 (NIH)
Record Dates: First submitted 2005-06-02; First posted 2005-06-03 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma; Recurrent Adult Brain Tumor
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Brain Neoplasms | interventions — Cilengitide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group I (high-dose cilengitide) 2000mg (Experimental): Preoperative Treatment: Patients receive high-dose cilengitide IV over 1 hour on days -8, -4, and -1. (High dose 2000mg)
  Resection: All patients undergo tumor resection on day 0.
  Postoperative Treatment: Beginning within 2 weeks after surgery, all patients receive high-dose cilengitide IV over 1 hour twice weekly for 4 weeks. Treatment repeats every 4 weeks for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: cilengitide; Procedure: therapeutic conventional surgery; Other: pharmacological study; Other: laboratory biomarker analysis
- Group II (low-dose cilengitide) 500mg (Experimental): Preoperative Treatment: Patients receive low-dose cilengitide IV over 1 hour on days -8, -4, and -1. (500mg)
  Resection: All patients undergo tumor resection on day 0.
  Postoperative Treatment: Beginning within 2 weeks after surgery, all patients receive high-dose cilengitide IV over 1 hour twice weekly for 4 weeks. Treatment repeats every 4 weeks for up to 24 courses in the absence of disease progression or unacceptable toxicity
  Interventions: Drug: cilengitide; Procedure: therapeutic conventional surgery; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: cilengitide — Given IV
  Other Names: EMD 121974
Procedure: therapeutic conventional surgery — Undergo tumor resection
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Cilengitide may stop the growth of glioblastoma multiforme by blocking blood flow to the tumor. Giving cilengitide before and after surgery may be an effective treatment for glioblastoma multiforme. This phase II trial is studying how well cilengitide works in treating patients who are undergoing surgery for recurrent or progressive glioblastoma multiforme.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the 6-month progression-free survival rate in operative patients with recurrent or progressive glioblastoma multiforme treated with cilengitide.

SECONDARY OBJECTIVES:

I. Determine the safety and toxicity of this drug in these patients.

OUTLINE: This is a multicenter study. Patients are randomized to 1 of 2 treatment groups for the preoperative treatment component.

Preoperative Treatment Group I: Patients receive high-dose cilengitide IV over 1 hour on days -8, -4, and -1.

Preoperative Treatment Group II: Patients receive low-dose cilengitide IV over 1 hour on days -8, -4, and -1.

Resection: All patients undergo tumor resection on day 0.

Postoperative Treatment: Beginning within 2 weeks after surgery, all patients receive high-dose cilengitide IV over 1 hour twice weekly for 4 weeks. Treatment repeats every 4 weeks for up to 24 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 44 patients (22 per preoperative treatment group) will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed intracranial glioblastoma multiforme (GBM)

  * Original diagnosis of low-grade glioma with subsequent histological confirmation of GBM allowed
  * Recurrent disease

    * Failed prior radiotherapy
* Must require a surgical procedure (gross total or near gross total resection) for tumor removal
* Performance status - Karnofsky 60-100%
* White Blood Count (WBC) ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10 g/dL (transfusion allowed)
* Serum glutamic oxaloacetic transaminase (SGOT) < 2 times upper limit of normal (ULN)
* Bilirubin < 2 times ULN
* Creatinine < 1.5 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for ≥ 2 weeks after study participation (for female patients) or for 3 months after study participation (for male patients)
* No other malignancy within the past 3 years except nonmelanoma skin cancer or carcinoma in situ of the cervix
* No active infection
* No other significant uncontrolled medical illness that would preclude study participation
* At least 3 weeks since prior interferon
* No prior cilengitide
* No other prior targeted antiangiogenic treatment (e.g., vatalanib, SU5416, or thalidomide)
* No concurrent anticancer immunotherapy
* No concurrent routine prophylactic filgrastim (G-CSF)
* At least 2 weeks since prior vincristine
* At least 3 weeks since prior procarbazine
* At least 6 weeks since prior nitrosoureas
* No concurrent anticancer chemotherapy
* At least 3 weeks since prior tamoxifen
* No concurrent anticancer hormonal therapy
* See Disease Characteristics
* At least 4 weeks since prior radiotherapy
* No concurrent anticancer radiotherapy
* Recovered from all prior therapies
* No more than 3 prior treatments for GBM (1 initial treatment; and treatment for 2 relapses)

  * For patients who received prior therapy for low-grade glioma, a subsequent surgical diagnosis of high-grade glioma is considered the first relapse
* At least 4 weeks since prior investigational agents
* At least 4 weeks since prior cytotoxic therapy
* At least 3 weeks since other prior non-cytotoxic therapy (e.g., isotretinoin), except radiosensitizers
* No other concurrent anticancer therapy
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-01; Primary Completion 2008-12 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Gilbert, Principal Investigator — North American Brain Tumor Consortium
Locations (1):
- North American Brain Tumor Consortium, Watertown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled from March 2005 through October 2006. Patients were recruited in the outpatient setting, however patients did need surgery for this study.
Groups:
- Low Dose 500mg Group 1: Preoperative Treatment: Patients receive low dose cilengitide 500mg IV over 1 hour on days -8, -4, and -1.
  Resection: All patients undergo tumor resection on day 0.
  Postoperative Treatment: Beginning within 2 weeks after surgery, all patients receive high-dose cilengitide 2000mg IV over 1 hour twice weekly for 4 weeks. Treatment repeats every 4 weeks for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  cilengitide: Given IV
  therapeutic conventional surgery: Undergo tumor resection
  pharmacological study: Correlative studies
  laboratory biomarker analysis: Correlative studies
- High Dose 2000mg Group 2: Preoperative Treatment: Patients receive high-dose cilengitide 2000mg IV over 1 hour on days -8, -4, and -1.
  Resection: All patients undergo tumor resection on day 0.
  Postoperative Treatment: Beginning within 2 weeks after surgery, all patients receive high-dose 2000mg cilengitide IV over 1 hour twice weekly for 4 weeks. Treatment repeats every 4 weeks for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  cilengitide: Given IV
  therapeutic conventional surgery: Undergo tumor resection
  pharmacological study: Correlative studies
  laboratory biomarker analysis: Correlative studies
Period: Overall Study
Arm/Group | Low Dose 500mg Group 1 | High Dose 2000mg Group 2
Started | 15 | 15
Completed | 13 | 13
Not Completed | 2 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — did not start treatment post-op | 1 | 2

BASELINE CHARACTERISTICS:
Population: 26 patients evaluated for toxicity and efficacy. 1 patient deemed ineligible and 3 patients did not re-start treatment post surgery.
Groups:
- Low Dose 500mg Group 1: Preoperative Treatment: Patients receive low dose 500mg cilengitide IV over 1 hour on days -8, -4, and -1.
  Resection: All patients undergo tumor resection on day 0.
  Postoperative Treatment: Beginning within 2 weeks after surgery, all patients receive high-dose 2000mg cilengitide IV over 1 hour twice weekly for 4 weeks. Treatment repeats every 4 weeks for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  cilengitide: Given IV
  therapeutic conventional surgery: Undergo tumor resection
  pharmacological study: Correlative studies
  laboratory biomarker analysis: Correlative studies
- High Dose 2000mg Group 2: Preoperative Treatment: Patients receive high-dose 2000mg cilengitide IV over 1 hour on days -8, -4, and -1.
  Resection: All patients undergo tumor resection on day 0.
  Postoperative Treatment: Beginning within 2 weeks after surgery, all patients receive high-dose 2000mg cilengitide IV over 1 hour twice weekly for 4 weeks. Treatment repeats every 4 weeks for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  cilengitide: Given IV
  therapeutic conventional surgery: Undergo tumor resection
  pharmacological study: Correlative studies
  laboratory biomarker analysis: Correlative studies
- Total: Total of all reporting groups
Arm/Group | Low Dose 500mg Group 1 | High Dose 2000mg Group 2 | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Median (Full Range); unit: years] | 51 [42 to 63] | 56 [42 to 68] | 55 [42 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 5 | 7 | 12
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 0 | 1 | 1
  White | 15 | 14 | 29
Histology - Glioblastoma [Number; unit: participants] | 15 | 15 | 30
Prior Chemotherapy [Number; unit: participants] | 15 | 15 | 30
Prior Immunotherapy [Number; unit: participants]
  Yes | 1 | 2 | 3
  No | 14 | 13 | 27
Prior Radiotherapy [Number; unit: participants] | 15 | 15 | 30
Prior Biopsy Only [Number; unit: participants]
  yes | 1 | 0 | 1
  no | 14 | 15 | 29

OUTCOME MEASURES:

1. Primary Outcome: 6m-Progression-free Survival
Description: progression within 6 months (26 weeks) of treatment
Time Frame: 6 months
Population: 6months progression free survival based on the post surgical treatment. All patients received 2000mg post surgery. The pre-surgery dose was used for correlative purposes only. All patients received surgery and the doses pre-surgery have no relation to the primary objective.
Measure: Number; unit: percent
Groups:
- Post-Operative Treatment 2000mg: Postoperative Treatment: Beginning within 2 weeks after surgery, all patients receive high-dose cilengitide IV over 1 hour twice weekly for 4 weeks. Treatment repeats every 4 weeks for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  cilengitide: Given IV
  pharmacological study: Correlative studies
Arm/Group | Post-Operative Treatment 2000mg
Number analyzed (Participants) | 26
percent | 12

2. Secondary Outcome: Changes in avb3 Integrin Expression on Tumor Cells and Endothelial Cells
Description: Will be performed between the untreated matched control tumor tissue and the tissue obtained from the post-treatment tumors using either a Fisher's Exact test or the Wilcoxon rank sum test depending on whether the assay provides a measurement or is yes/no.
Time Frame: Baseline and time of surgery
Population: Molecular analyses evaluating alterations after cilengitide treatments were planned as a component of this clinical trial, unfortunately, the majority of tumor samples were too small to do both measures of drug and molecular analysis or the sample was inadequate for both after removal of areas of necrosis and gliosis
Groups:
- Group I Pre-op (Low-dose Cilengitide) 500mg: Preoperative Treatment: Patients receive low-dose cilengitide IV over 1 hour on days -8, -4, and -1. (low dose 500mg)
  Resection: All patients undergo tumor resection on day 0.
  cilengitide: Given IV therapeutic conventional surgery: Undergo tumor resection
  laboratory biomarker analysis: Correlative studies
- Group II Pre-op (High-dose Cilengitide) 2000mg: Preoperative Treatment: Patients receive high-dose cilengitide IV over 1 hour on days -8, -4, and -1. (2000mg)
  Resection: All patients undergo tumor resection on day 0.
  cilengitide: Given IV therapeutic conventional surgery: Undergo tumor resection laboratory biomarker analysis: Correlative studies
Arm/Group | Group I Pre-op (Low-dose Cilengitide) 500mg | Group II Pre-op (High-dose Cilengitide) 2000mg
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Changes in Vitronectin Expression
Description: as for outcome 2
Time Frame: Baseline and time of surgery
Population: Molecular analyses evaluating alterations planned, unfortunately, majority of tumor samples were too small to do both measures of drug and molecular analysis or sample was inadequate for both after removal of areas of necrosis and gliosis
Arm/Group | Group I Pre-op (Low-dose Cilengitide) 500mg | Group II Pre-op (High-dose Cilengitide) 2000mg
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Changes in Tumor Cell Apoptosis
Description: as for outcome 2
Time Frame: Baseline and time of surgery
Population: as for outcome 3
Groups:
- Group II Pre-op (High-dose Cilengitide) 2000mg: Preoperative Treatment: Patients receive low-dose cilengitide IV over 1 hour on days -8, -4, and -1. (low dose 500mg)
  Resection: All patients undergo tumor resection on day 0.
  cilengitide: Given IV therapeutic conventional surgery: Undergo tumor resection
  laboratory biomarker analysis: Correlative studies
Arm/Group | Group I Pre-op (Low-dose Cilengitide) 500mg | Group II Pre-op (High-dose Cilengitide) 2000mg
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Changes in Tumor Cell Proliferation
Description: as for outcome 2
Time Frame: Baseline and time of surgery
Population: as for outcome 3
Arm/Group | Group I Pre-op (Low-dose Cilengitide) 500mg | Group II Pre-op (High-dose Cilengitide) 2000mg
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Changes in Endothelial Cell Apoptosis
Description: as for outcome 2
Time Frame: Baseline and up to 4 years
Population: as for outcome 3
Arm/Group | Group II Pre-op (High-dose Cilengitide) 2000mg | Group I Pre-op (Low-dose Cilengitide) 500mg
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Plasma Concentration of EMD 121974
Description: 24 hour post dose concentration plasma, at time of resection
Time Frame: 24 hour post concentration
Population: 6 of 8 and 7 of 11 plasma samples at the 500mg and 2000mg dose level respectively, were below the lower level of quantitation (LLOQ) Of the 15 samples in the low dose group only 8 were evaluable and 11 of the 15 for the high dose group. Samples were either damaged or too small for analysis.
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Group I (Low-dose Cilengitide) 500mg: Preoperative Treatment: Patients receive low-dose cilengitide IV over 1 hour on days -8, -4, and -1. (High dose 2000mg)
  Resection: All patients undergo tumor resection on day 0.
  Postoperative Treatment: Beginning within 2 weeks after surgery, all patients receive 2000mg high-dose cilengitide IV over 1 hour twice weekly for 4 weeks. Treatment repeats every 4 weeks for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  cilengitide: Given IV
  therapeutic conventional surgery: Undergo tumor resection
  pharmacological study: Correlative studies
  laboratory biomarker analysis: Correlative studies
- Group II High-dose Cilengitide) 2000mg: Preoperative Treatment: Patients receive high-dose cilengitide IV over 1 hour on days -8, -4, and -1. (2000mg)
  Resection: All patients undergo tumor resection on day 0.
  Postoperative Treatment: Beginning within 2 weeks after surgery, all patients receive high-dose 2000mg cilengitide IV over 1 hour twice weekly for 4 weeks. Treatment repeats every 4 weeks for up to 24 courses in the absence of disease progression or unacceptable toxicity
  cilengitide: Given IV
  therapeutic conventional surgery: Undergo tumor resection
  pharmacological study: Correlative studies
  laboratory biomarker analysis: Correlative studies
Arm/Group | Group I (Low-dose Cilengitide) 500mg | Group II High-dose Cilengitide) 2000mg
Number analyzed (Participants) | 8 | 11
ng/ml | 333 (16.97) | 386 (184)

8. Secondary Outcome: Tumor Tissue Concentrations
Description: a section of tumor of approximately 500mg will be snap frozen (immediately prepared and frozen) once removed from brain for analysis of the drug concentration in contrast -enhancing tumor.
Time Frame: at time of surgery
Population: 8 500mg dose tissue samples and 10 2000mg dose tissue samples were either too small or had large areas of necrosis and gliosis to do analysis/evaluation
Measure: Mean (Standard Deviation); unit: ng/g
Groups:
- Group I (Low-dose Cilengitide) 500mg: Preoperative Treatment: Patients receive low-dose cilengitide IV over 1 hour on days -8, -4, and -1. (low dose 500mg)
  Resection: All patients undergo tumor resection on day 0.
  Postoperative Treatment: Beginning within 2 weeks after surgery, all patients receive high-dose 2000mg cilengitide IV over 1 hour twice weekly for 4 weeks. Treatment repeats every 4 weeks for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  cilengitide: Given IV
  therapeutic conventional surgery: Undergo tumor resection
  pharmacological study: Correlative studies
  laboratory biomarker analysis: Correlative studies
- Group II (High-dose Cilengitide) 2000mg: Preoperative Treatment: Patients receive high-dose cilengitide IV over 1 hour on days -8, -4, and -1. (2000mg)
  Resection: All patients undergo tumor resection on day 0.
  Postoperative Treatment: Beginning within 2 weeks after surgery, all patients receive high-dose 2000mg cilengitide IV over 1 hour twice weekly for 4 weeks. Treatment repeats every 4 weeks for up to 24 courses in the absence of disease progression or unacceptable toxicity
  cilengitide: Given IV
  therapeutic conventional surgery: Undergo tumor resection
  pharmacological study: Correlative studies
  laboratory biomarker analysis: Correlative studies
Arm/Group | Group I (Low-dose Cilengitide) 500mg | Group II (High-dose Cilengitide) 2000mg
Number analyzed (Participants) | 7 | 5
ng/g | 919 (1235) | 1413 (1335)

9. Other Pre Specified Outcome: Overall Progression Free Survival
Description: Kaplan-meier curve
Time Frame: 1 year
Population: Overall survival based on the post surgical treatment. All patients received 2000mg post surgery. The pre-surgery dose was used for correlative purposes only. All patients received surgery and the doses pre-surgery have no relation to the this objective.
Measure: Median (95% Confidence Interval); unit: weeks
Groups:
- Post-Operative Treatment 2000mg: Postoperative Treatment: Beginning within 2 weeks after surgery, all patients receive high-dose 2000mg cilengitide IV over 1 hour twice weekly for 4 weeks. Treatment repeats every 4 weeks for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  cilengitide: Given IV
  therapeutic conventional surgery: Undergo tumor resection
  pharmacological study: Correlative studies
  laboratory biomarker analysis: Correlative studies
Arm/Group | Post-Operative Treatment 2000mg
Number analyzed (Participants) | 26
weeks | 8 [4 to 16]

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Post-Operative 2000mg: Postoperative Treatment: Beginning within 2 weeks after surgery, all patients receive high-dose 2000mg cilengitide IV over 1 hour twice weekly for 4 weeks. Treatment repeats every 4 weeks for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  cilengitide: Given IV
  therapeutic conventional surgery: Undergo tumor resection
  pharmacological study: Correlative studies
  laboratory biomarker analysis: Correlative studies
Arm/Group | Post-Operative 2000mg
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 26/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Post-Operative 2000mg (N=26)
Alanine aminotransferase (Investigations) | 2 (2)
anorexia (Metabolism and nutrition disorders) | 2 (2)
bruising (Injury, poisoning and procedural complications) | 2 (2)
diarrhea (Gastrointestinal disorders) | 2 (2)
fatigue (General disorders) | 8 (8)
hemoglobin (Investigations) | 8 (8)
hyperglycemia (Metabolism and nutrition disorders) | 3 (3)
hyponatremia (Metabolism and nutrition disorders) | 2 (2)
hypoalbuminemia (Metabolism and nutrition disorders) | 3 (3)
leukocytes (Blood and lymphatic system disorders) | 10 (10)
lymphopenia (Blood and lymphatic system disorders) | 11 (11)
nausea (Gastrointestinal disorders) | 3 (3)
neutrophils (Investigations) | 3 (3)
platelets (Investigations) | 6 (6)

LIMITATIONS AND CAVEATS:
Study closed early due to slow accrual. Molecular analyses evaluating alterations were planned for the study, unfortunately, majority of tumor samples were too small to do analysis and also there were unforeseen freezer issues.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less